CLINICAL TRIAL: NCT03542643
Title: A Double-blind Randomised Controlled Trial of N-3 PUFAs in Children With Attention Deficit Hyperactivity Disorder
Brief Title: Omega-3 Polyunsaturated Fatty Acids in Youth With ADHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMUH104-REC2-058
Record Dates: First submitted 2018-05-20; First posted 2018-05-31 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Attention Deficit Hyperactivity Disorder; ADHD
Keywords: ADHD; n-3 polyunsaturated fatty acids; children; adolescents
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-3 polyunsaturated fatty acids (Active Comparator): n-3 polyunsaturated fatty acids dosage of 1g of Eicosapentaenoic acid(EPA)
  Interventions: Dietary Supplement: n-3 Polyunsaturated fatty acid
- Placebo (Placebo Comparator): olive oil ethyl esters
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: n-3 Polyunsaturated fatty acid — 1g of Eicosapentaenoic acid (EPA)
  Arms: N-3 polyunsaturated fatty acids
Dietary Supplement: Placebo — Olive oil ethyl esters
  Arms: Placebo

SUMMARY:
N-3 polyunsaturated fatty acids(N-3 PUFAs) is important in balancing the immune function and crucial for the developing brain. Deficiency in n-3 PUFAs might be linked to the poor cognitive performances resulting in inattention and hyperactivity in youth with attention deficit hyperactivity disorder (ADHD). N-3 PUFAs appears to be a promising treatment that is safe, beneficial to youth with ADHD. In this proposal, investigators aim the test the hypothesis that n-3 polyunsaturated fatty acids will be more effective than placebo in improving cognitive function in youth with ADHD after 12 weeks of intervention.

DETAILED DESCRIPTION:
This is a 1-year study and a randomized, double-blind, and placebo controlled Clinical the study. investigators plan to enrol 100 subjects from Child and Adolescent Psychiatry Outpatient Clinic of China Medical University Hospital.Participants will be randomized into omega-3 polyunsaturated fatty acids or placebo group.The intervention period is 12 weeks. Evaluation of the cognitive function ( using Continuous Performance Test 3rd Edition ) of the subjects who are enrolled into the study will take place at baseline and after the 12th week. The symptom severity of ADHD will be measured with Swanson, Nolan, Pelham Questionnaire (SNAP-IV) at baseline, 2,4,8, and 12 weeks. The plasma level of n-3 polyunsaturated fatty acids, blood and salivary inflammatory markers will also be measured at the beginning and at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* DSM-5 diagnosed ADHD
* Age 6-18 years old at time of enrolment
* Conner's rating scares (CPRS) with scores >= 2 standard deviations
* drug native or no medication use for past 6 months
* Signed informed consent

Exclusion Criteria:

* Intelligence quotient <70
* Comorbid other psychiatric disorders, such as autism spectrum disorders, anxiety disorders, conduct disorders, schizophrenia, major depressive disorders and bipolar spectrum disorders
* Comorbid physical disorders, such as thyroid dysfunction, cerebral palsy
* Current using omega-3 supplements
* Allergy to omega-3

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 105 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Changes in Continuous Performance Test Raw Scores at 12 weeks | Week 0 and Week 12
  Correct Detection: This indicates the number of times the client responded to the target stimulus. Higher rates of correct detections indicate better attentional capacity.
  Reaction times: This measures the amount of time between the presentation of the stimulus and the client's response.
  Omission errors: This indicates the number of times the target was presented, but the client did not respond/click the mouse. High omission rates indicate that the subject is either not paying attention (distractibility) to stimuli or has a sluggish response.
  Commission errors: This score indicates the number of times the client responded but no target was presented. A fast reaction time and high commission error rate points to difficulties with impulsivity. A slow reaction time with high commission and omission errors, indicates inattention in general.

SECONDARY OUTCOMES:
Changes in SNAP-IV Scores for Inattention, Hyperactivity and Total ADHD Symptom Severity | Week 0, 2,4,8,12
  Inattention: items 1-9 Hyperactivity: items 10-18 Total ADHD: items 1-18 the greater the scores on SNAP-IV indicate the greater the severity of ADHD symptoms

OTHER OUTCOMES:
Changes in Blood PUFAs levels at 12 Weeks | Week 0 and Week 12
  measurement of blood PUFAs levels
Changes in Blood Inflammatory Markers at 12 Weeks | Week 0 and Week 12
  measurements of blood inflammatory markers
Changes in Salivary Cortisol at 12 Weeks | Week 0 and Week 12
  measurements of salivary cortisol

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taiwan

REFERENCES:
- [Derived] Gillies D, Leach MJ, Perez Algorta G. Polyunsaturated fatty acids (PUFA) for attention deficit hyperactivity disorder (ADHD) in children and adolescents. Cochrane Database Syst Rev. 2023 Apr 14;4(4):CD007986. doi: 10.1002/14651858.CD007986.pub3. PMID 37058600